CLINICAL TRIAL: NCT06463769
Title: "Impact of Diet on the Microbiome-Immune-Brain Axis in Parkinson's Disease" as Part of the Collaborative Research Center 1697 "Targeting the Microbiome-Immune-Brain Interaction in Neurodegeneration"
Brief Title: Impact of Diet on the Microbiome-Immune-Brain Axis in Parkinson's Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kiel (Other)
Collaborators: University Hospital Schleswig-Holstein (Other)
Responsible Party: Principal Investigator, Prof. Dr. Dr. Anja Bosy-Westphal, Head of the Department of Human Nutrition, Kiel University, University of Kiel
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRC1697-C04
Record Dates: First submitted 2024-06-05; First posted 2024-06-18 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Parkinson Disease
Keywords: New Nordic Diet; Parkinson's Disease; Microbiome-Immune-Brain axis
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Arm 1: Patients with prodromal PD receiving nutritional intervention Arm 2: Patients with clinical PD receiving nutritional intervention Arm 3: Patients with clinical PD receiving standard of care (control)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patients with prodromal PD on New Nordic LPF-diet (intervention) (Experimental): Patients with prodromal PD will take part in an 8-week patient-centered intervention program on a predominantly plant-based New Nordic LPF-Diet.
  Interventions: Behavioral: 8 week predominantly plant-based New Nordic LPF-diet program; Behavioral: maintenance of the predominantly plant-based New Nordic LPF-diet
- Patients with clinical PD on New Nordic LPF-diet (intervention) (Experimental): Patients with clinical PD will take part in an 8-week patient-centered intervention program on a predominantly plant-based New Nordic LPF-Diet. Patients with clinical PD will be randomized to intervention or control group.
  Interventions: Behavioral: 8 week predominantly plant-based New Nordic LPF-diet program; Behavioral: maintenance of the predominantly plant-based New Nordic LPF-diet
- Patients with clinical PD receiving standard of care (control) (No Intervention): Patients with clinical PD will receive standard of care information on a healthy diet and serve as control. Patients with clinical PD will be randomized to intervention or control group.

INTERVENTIONS:
Behavioral: 8 week predominantly plant-based New Nordic LPF-diet program — An 8-week patient-centered dietary intervention program will be implemented to maintain a predominantly plant-based New Nordic LPF-Diet.
  Arms: Patients with clinical PD on New Nordic LPF-diet (intervention); Patients with prodromal PD on New Nordic LPF-diet (intervention)
Behavioral: maintenance of the predominantly plant-based New Nordic LPF-diet — Follow-up of long-term adherence to the diet at one and six months after completion of the intervention program.
  Arms: Patients with clinical PD on New Nordic LPF-diet (intervention); Patients with prodromal PD on New Nordic LPF-diet (intervention)

SUMMARY:
Habitual adherence to a predominantly plant-based diet, rich in low-processed food (LPF) has been associated with a reduced risk for development and slower progression of Parkinson's Disease (PD). This could be due to neuroprotective effects by modulation of the gut microbiota and decreased neuronal and metabolic inflammation. So far, the effect of a predominantly plant-based LPF-diet on the microbiome-immune-brain axis in patients with PD remains unknown. In addition, the influence of dietetic measures on the gut microbiome is variable and may depend on (long-term) adherence as well as on PD-specific factors and lifestyle.

The investigators hypothesize that compared to an average German diet, the predominantly plant-based New Nordic LPF-diet, as a culturally adapted diet, which is rich in fermentable fiber and phytochemicals, will have beneficial effects on the gut microbiome of patients with PD by increasing the abundance of short-chain fatty acid (SCFA)-producing bacteria (primary outcome) and will improve gut motility, metabolic resilience, and inflammation (secondary outcomes). Furthermore, the investigators postulate that a patient-centered dietary intervention program, including a multifaceted patient education and supported by a web-application, will lead to high adherence as a key determinant of long-term changes in the gut microbiome. This dietary intervention will be accepted by patients as a low-threshold treatment that balances personal benefits, therapeutic barriers and ethical concerns of early risk disclosure in PD.

DETAILED DESCRIPTION:
In a pilot-intervention study, our project will:

* develop a practical, low-threshold diet intervention for patients with prodromal and clinical PD. Adherence will be promoted (i) by a patient-oriented approach, (ii) by implementation of the predominantly plant-based New Nordic LPF-diet that is scientifically-based, culturally adapted, sustainable and culinary and (iii) by an innovative web-application.
* investigate the acute effects of the predominantly plant-based New Nordic LPF -diet on the microbiome (abundance of SCFA-producing bacteria), gastrointestinal motility, inflammation as well as metabolic and Parkinson-specific clinical outcomes in individuals with prodromal and clinical PD.
* investigate potential determinants of long-term changes in the gut microbiome (e.g. dietary adherence, gastrointestinal motility, meal timing and frequency), and factors associated with a high adherence (e.g. acceptance of diet as therapeutic intervention in the prodromal phase, health-related quality of life).

The patient-centered intervention program will be tailored to individual needs and preferences of individuals with prodromal and clinical PD. It will be designed to impart knowledge (e.g. on sustainability and health effects) and food literacy (e.g. food merchandize and culinary skills) in group meetings and culinary medicine workshops. Recipe suggestions and shopping guides will consider individual abilities and needs and a web-application is used for information, increasing self-efficacy, motivation, and monitoring. To ensure an easy integration of the diet into everyday life, partners will be included in the program, if applicable. Moreover, cultural preferences as well as financial resources will be considered. Regular feedback using statistics on nutrient intake and overall progress will be implemented to encourage adherence.

ELIGIBILITY:
Inclusion Criteria:

* patients with probable prodromal PD (according to predefined criteria)
* patients with clinical PD with slight to moderate disease severity (Hoehn & Yahr 1-2.5)
* habitual Western Diet (≥30% of energy intake from ultra-processed food)

Exclusion Criteria:

* current adherence to a plant-based diet
* food allergies or intolerances
* significant diseases of the gastrointestinal system (e.g. celiac disease) or central nervous system, diabetes mellitus
* underweight (BMI <18.5 kg/m2)
* active smoking
* expected changes in medication or antibiotic treatment during the intervention

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
abundance of key SCFA-producing gut bacteria | pre vs. post intervention (8 weeks) + pre intervention vs. follow-up 6 months after completion of intervention
  analysis of stool samples

SECONDARY OUTCOMES:
systemic inflammation markers | pre vs. post intervention (8 weeks) + pre intervention vs. follow-up 6 months after completion of intervention
  hsCRP and IL-6 in serum
metabolic resilience | pre vs. post intervention (8 weeks)
  modeling of one parameter (metabolic resilience) including information on postprandial glucose, insulin, triglycerides and NEFA following a mixed meal tolerance test
gastrointestinal peptide-hormones | pre vs. post intervention (8 weeks)
  ghrelin, GLP-1, PYY
energy balance | pre vs. post intervention (8 weeks) + pre intervention vs. follow-up 6 months after completion of intervention
  changes in body weight
energy partitioning | pre vs. post intervention (8 weeks) + pre intervention vs. follow-up 6 months after completion of intervention
  changes in body composition

OTHER OUTCOMES:
clinical motor symptoms | pre vs. post intervention (8 weeks) + pre intervention vs. follow-up 6 months after completion of intervention
  clinical examination
clinical non-motor symptoms | pre vs. post intervention (8 weeks) + pre intervention vs. follow-up 6 months after completion of intervention
  clinical examination
gastric emptying | pre vs. post intervention (8 weeks) + pre intervention vs. follow-up 6 months after completion of intervention
  13C-breath test
gastrointestinal transit time | pre vs. post intervention (8 weeks) + pre intervention vs. follow-up 6 months after completion of intervention
  using a test meal with food colouring and the time to colour appearance in stool
gut motility | pre vs. post intervention (8 weeks) + pre intervention vs. follow-up 6 months after completion of intervention
  functional visceral MRI
dietary adherence via serum markers | pre vs. post intervention (8 weeks) + pre intervention vs. follow-up 6 months after completion of intervention
  serum carotinoid and Trimethylamine oxid-levels will be combined and tertiles will be formed
dietary adherence via healthy Nordic food Index | pre vs. post intervention (8 weeks) + pre intervention vs. follow-up 6 months after completion of intervention
  healthy Nordic food Index using data from a food frequency questionnaire
food literacy effectiveness | pre vs. post intervention (8 weeks) + pre intervention vs. follow-up 6 months after completion of intervention
  self-perceived food literacy scale (questionnaire)
patient acceptance | pre vs. post intervention (8 weeks) + pre intervention vs. follow-up 6 months after completion of intervention
  Parkinson's Disease Questionnaire (PDQ-39)
patient quality of life | pre vs. post intervention (8 weeks) + pre intervention vs. follow-up 6 months after completion of intervention
  Ways of Coping Questionnaire (WCQ)

CONTACTS AND LOCATIONS:
Overall Officials: Anja Bosy-Westphal, PhD, MD, Principal Investigator — Kiel University; Eva Schäffer, MD, Principal Investigator — Kiel University, University Hospital Schleswig-Holstein
Locations (2):
- Germany (2):
  - Institute of Human Nutrition, Kiel
  - Kiel University, University Hospital Schleswig-Holstein, Kiel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aho VTE, Houser MC, Pereira PAB, Chang J, Rudi K, Paulin L, Hertzberg V, Auvinen P, Tansey MG, Scheperjans F. Relationships of gut microbiota, short-chain fatty acids, inflammation, and the gut barrier in Parkinson's disease. Mol Neurodegener. 2021 Feb 8;16(1):6. doi: 10.1186/s13024-021-00427-6. PMID 33557896
- [Background] Solch RJ, Aigbogun JO, Voyiadjis AG, Talkington GM, Darensbourg RM, O'Connell S, Pickett KM, Perez SR, Maraganore DM. Mediterranean diet adherence, gut microbiota, and Alzheimer's or Parkinson's disease risk: A systematic review. J Neurol Sci. 2022 Mar 15;434:120166. doi: 10.1016/j.jns.2022.120166. Epub 2022 Jan 26. PMID 35144237
- [Background] Maraki MI, Yannakoulia M, Stamelou M, Stefanis L, Xiromerisiou G, Kosmidis MH, Dardiotis E, Hadjigeorgiou GM, Sakka P, Anastasiou CA, Simopoulou E, Scarmeas N. Mediterranean diet adherence is related to reduced probability of prodromal Parkinson's disease. Mov Disord. 2019 Jan;34(1):48-57. doi: 10.1002/mds.27489. Epub 2018 Oct 10. PMID 30306634